CLINICAL TRIAL: NCT03584451
Title: Randomized, Clinical Survey for Evaluating the Effect of Rehabilitation Sport on Patients Who Underwent Total Hip Arthroplasty (THA)
Brief Title: Evaluation of the Effect of Rehabilitation Sport After Total Hip Arthroplasty (THA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rehasport after THA
Record Dates: First submitted 2018-06-04; First posted 2018-07-12 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Total Hip Arthroplasty; Osteoarthritis, Hip; Sports Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with rehabilitation sport (Active Comparator): rehabilitation sport over 52 weeks after THA, start 6 weeks postoperatively
  Interventions: Behavioral: rehabilitation sport
- without rehabilitation sport (No Intervention): no further rehabilitation program after THA

INTERVENTIONS:
Behavioral: rehabilitation sport — rehabilitation Sport over 52 weeks after THA, start 6 weeks postoperatively
  Arms: with rehabilitation sport

SUMMARY:
160 patients who received a total hip arthroplasty (THA) were included and randomized to receive specific rehabilitation sport (RS) or not (control) in addition to a conventional rehabilitation program. Upon completion of the rehabilitation phase 6 weeks, 6 months and 12 months after surgery sports medical measurements have been performed. Strength abilities of the hip muscles were tested with isokinetic dynamometry, postural control with a force measuring platform and endurance via lactate measurements.

DETAILED DESCRIPTION:
In Germany, rehabilitation sport (RS) is a reimbursed postoperative measure in order to support socio-professional reintegration and self-help.

160 patients who received a primary total hip arthroplasty (THA) were included and randomized to receive specific RS or not (control) in addition to a conventional rehabilitation program. Upon completion of the rehabilitation phase 6 weeks, 6 months and 12 months after surgery sports medical measurements have been performed. Strength abilities of the hip muscles were tested with isokinetic dynamometry, postural control with a force measuring platform and endurance via lactate measurements. The goal of the study was to prospectively randomized evaluate the effect of RS on hip-related muscular strength, endurance and postural stability on patients who underwent THA.

ELIGIBILITY:
Inclusion Criteria:

* non-complicated THA
* written informed consent

Exclusion Criteria:

* complicated THA
* partial weight-bearing after surgery
* cardial comorbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
hip-related muscular strength | change from baseline (6 weeks) at 6 months after THA
  hip-related muscular strength measured with isokinetic dynamometry

SECONDARY OUTCOMES:
Hip pain - WOMAC | change from 6 months to 12 months after THA
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscore (worst=0, best=100)
Physical function hip - WOMAC | change from 6 months to 12 months after THA
  WOMAC Total Score (worst=0, best=100)
Physical function hip - HHS | change from 6 months to 12 months after THA
  Harris-Hip-Score (worst=0, best=100)
Physical Activity | change from 6 months to 12 months after THA
  University of California, Los Angeles (UCLA) Activity Scale (worst=1, best=10)
health related Quality of life | change from 6 months to 12 months after THA
  EuroQol in 5 dimensions (EQ-5D) Index (worst=0, best=1), EQ-VAS (worst=0, best=100)
Hip pain | change from 6 months to 12 months after THA
  Visual Analogue Scale (worst=0, best=10)
cardiovascular endurance | change from baseline (6 weeks) at 6 months after THA
  cardiovascular endurance via lactate measurements
cardiovascular endurance | change from baseline (6 weeks) at 12 months after THA
  cardiovascular endurance via lactate measurements
postural control | change from baseline (6 weeks) at 6 months after THA
  postural control with a force measuring platform
postural control | change from baseline (6 weeks) at 12 months after THA
  postural control with a force measuring platform
hip-related muscular strength | change from baseline (6 weeks) at 12 months after THA
  hip-related muscular strength measured with isokinetic dynamometry

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD